CLINICAL TRIAL: NCT01039584
Title: A Randomized Study Evaluating the Therapeutic Equivalence and Safety of Butoconazole Nitrate Vaginal Cream, 2% and Gynazole 1 (Butoconazole Nitrate) Vaginal Cream, 2%, Against a Vehicle Control in the Treatment of Vulvovaginal Candidiasis
Brief Title: A Randomized Study Evaluating the Therapeutic Equivalence of Two Butoconazole Nitrate Vaginal Cream, 2% Formulations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Padagis LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRG-710
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Results first posted 2013-01-21 (Estimated); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Vulvovaginal Candidiasis
Keywords: bioequivalence; butoconazole; vulvovaginal; candidiasis
MeSH Terms: conditions — Candidiasis, Vulvovaginal; Candidiasis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): vehicle of the test product; applied intravaginally once within 48 hours of randomization
  Interventions: Drug: Placebo
- Test Product (Experimental): Butoconazole Nitrate Vaginal Cream; applied intravaginally once within 48 hours of randomization
  Interventions: Drug: Butoconazole Nitrate Vaginal Cream
- Reference Product (Active Comparator): Gynazole 1 Vaginal Cream; applied intravaginally once within 48 hours of randomization
  Interventions: Drug: Gynazole 1 vaginal cream

INTERVENTIONS:
Drug: Butoconazole Nitrate Vaginal Cream — vaginal cream
  Arms: Test Product
Drug: Placebo — vaginal cream
  Other Names: vehicle of the test product
  Arms: Placebo
Drug: Gynazole 1 vaginal cream — vaginal cream
  Other Names: Gynazole 1
  Arms: Reference Product

SUMMARY:
This was a study that compared the efficacy and safety of a generic butoconazole nitrate vaginal cream, 2% to Gynazole-1 (butoconazole nitrate) Vaginal Cream, 2% in the treatment of vulvovaginal candidiasis caused by Candida species.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects, at least 18 years of age
* Presented with symptomatic vulvovaginitis consistent with a diagnosis of moniliasis
* Signed and dated informed consent

Exclusion Criteria:

* Were pregnant, nursing, or planning a pregnancy within the study participation period
* Had evidence of any bacterial, viral, or protozoal infection
* Had hypersensitivity or allergy to the imidazoles, their analogues, and/or any of the Test Product ingredients
* Had any medical condition, or used any medication which, in the opinion of the investigator, could have interfered with the conduct of the study

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 611 (Actual)
Dates: Start 2008-02; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PharmaNet, Inc. (PharmaNet), Charlotte, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Product: Butoconazole Nitrate Vaginal Cream
  Butoconazole Nitrate Vaginal Cream : vaginal cream
- Reference Product: Gynazole 1 Vaginal Cream
  Gynazole 1 vaginal cream : vaginal cream
- Placebo: vehicle of the test product
  Placebo : vaginal cream
Period: Overall Study
Arm/Group | Test Product | Reference Product | Placebo
Started | 246 | 243 | 122
Completed | 143 | 146 | 65
Not Completed | 103 | 97 | 57
Not completed — Withdrawal by Subject | 4 | 2 | 1
Not completed — Protocol Violation | 10 | 4 | 6
Not completed — Lost to Follow-up | 5 | 3 | 4
Not completed — Negative Baseline culture for Candida | 59 | 59 | 24
Not completed — Lack of Efficacy | 7 | 6 | 10
Not completed — other | 1 | 3 | 1
Not completed — Pap smear with significant pathology | 10 | 10 | 3
Not completed — Positive for Chlamydia or gonorrhea | 7 | 10 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Product | Reference Product | Placebo | Total
Number analyzed (Participants) | 246 | 243 | 122 | 611
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 5 | 4 | 17
  Between 18 and 65 years | 236 | 238 | 117 | 591
  >=65 years | 2 | 0 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.1 (10.29) | 32.1 (10.02) | 33.3 (11.15) | 32.3 (10.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 246 | 243 | 122 | 611
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 108 | 107 | 54 | 269
  Central America | 54 | 53 | 26 | 133
  South America | 84 | 83 | 42 | 209

OUTCOME MEASURES:

1. Primary Outcome: The Test of Equivalence Between the Test and Reference Products Was Based on the Therapeutic Cure Rates at Visit 3/Test-of-Cure.
Description: Therapeutic cure is defined as both the mycologically-proven eradication of infection caused by Candida species (mycological cure) and evidence of clinical success (clinical cure)
Time Frame: Visit 3: Day 22-31
Population: per-protocol
Measure: Number; unit: participants
Arm/Group | Test Product | Reference Product | Placebo
Number analyzed (Participants) | 137 | 133 | 67
participants | 73 | 73 | 16
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — The primary efficacy measure was the proportion of subjects with therapeutic cure at Visit 3/Test-of-Cure. Therapeutic cure was defined as having both a mycological cure and a clinical cure; Wald's method; Yates continuity correction = 1.5, 90% CI 2-sided [-9.1 to 12.3]

2. Secondary Outcome: Clinical Cure
Description: Clinical cure (clinical success) was defined as follows:
  1. All signs or symptoms with a score of 1 (mild) or 2 (moderate) at Visit 1/Baseline had a score of 0 (absent) at Visit 3/Test-of-Cure, or all signs or symptoms with a score of 3 (severe) at Visit 1/Baseline had a score of 0 (absent) or 1 (mild) at Visit 3/Test-of-Cure
  2. A new sign or symptoms was observed at Visit 3/Test-of-Cure that was not present at entry and was determined by the investigator to not be related to VVC (if related, the subject was considered a failure; if not related, the subject could have been considered a cure)
  3. The subject did not require additional vulvovaginal or systemic antifungal therapy
  4. The subject did not use any topical drug therapy other than the study medication for the treatment of vulvovaginal irritation and/or pruritus, such as topical analgesics or corticosteroid products
Time Frame: Visit 3: Day 22-31
Population: per-protocol
Measure: Number; unit: participants
Arm/Group | Test Product | Reference Product | Placebo
Number analyzed (Participants) | 137 | 133 | 67
participants | 91 | 92 | 32
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — The efficacy measure was the proportion of subjects with clinicl cure at Visit 3/Test-of-Cure; Wald's method; Yates continuity correction = 1.5, 90% CI 2-sided [-7.3 to 12.8]

3. Secondary Outcome: Mycological Cure
Description: Mycological cure was defined as a negative mycological culture (no growth)
Time Frame: Visit 3: Day 22-31
Measure: Number; unit: participants
Arm/Group | Test Product | Reference Product | Placebo
Number analyzed (Participants) | 137 | 133 | 67
participants | 83 | 79 | 18
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — The efficacy measure was the proportion of subjects with mycological cure at Visit 3/Test-of-Cure; p = 0.05, Wald's method; Yates continuity correction = 1.5, 90% CI 2-sided [-11.7 to 9.4]

ADVERSE EVENTS:
Time Frame: From the signing of informed consent to 30 days post subject participation.
Arm/Group | Test Product | Reference Product | Placebo
Serious Adverse Events (participants affected / at risk) | 0/246 | 0/243 | 0/122
Other Adverse Events (participants affected / at risk) | 0/246 | 0/243 | 0/122

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other